CLINICAL TRIAL: NCT04556279
Title: Investigating Salt Taste Threshold in Patients Being Investigated for Primary Hyperaldosteronism Before and After Treatment.
Acronym: AldoSalt
Status: Withdrawn | Type: Observational
Why Stopped: Researcher's Decision
Sponsor: Imperial College London (Other)
Collaborators: Institute of Neuroscience and Medicine, Julich, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20HH6283
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hyperaldosteronism; Primary; Hypertension; Salt; Excess; Appetite Disorders
MeSH Terms: conditions — Hyperaldosteronism; Hypertension; Feeding and Eating Disorders | interventions — Adrenalectomy; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- hyperaldosteronism surgical treatment: Hypertensive patients with primary hypersldosteronism, treated with surgery
  Interventions: Procedure: adrenalectomy
- hyperaldosteronism medical treatment: Hypertensive patients with primary hypersldosteronism, treated with aldosterone blockade.
  Interventions: Drug: Aldosterone Antagonist
- hypertensive control: Hypertensive patients shown not to have primary hyperaldosteronism

INTERVENTIONS:
Procedure: adrenalectomy — Surgical removal of an adrenal gland containing an aldosterone secreting adenoma.
  Other Names: aldosterone blockade
  Groups: hyperaldosteronism surgical treatment
Drug: Aldosterone Antagonist — Medical treatment of primary hyperaldosteronism.
  Groups: hyperaldosteronism medical treatment

SUMMARY:
This study looks at how hypertensive patients, with high levels of aldosterone (hyperaldosteronism) differ from hypertensive patients without hyperaldosteronism with regards to markers of salt appetite. It also looks at how salt appetite changes after treatment of hyperaldosteronism. Salt makes food taste good and when our bodies need salt our brains make us like salty food even more. A high salt diet contributes to hypertension and a low salt diet is an important aspect of the treatment of hypertension. Unfortunately patients find it difficult to adhere to a low salt diet. Aldosterone is produced by the adrenal glands, its release is stimulated by a salt need and it has been shown, in rodent models, to activate pathways in the brain which drive a salt appetite. Mice with enhanced activity of the aldosterone pathway in the brain become hypertensive due to increased salt intake. Hyperaldosteronism, in humans, results in hypertension. The contribution of salt appetite, as opposed to the effect of aldosterone on the kidney's retention of salt and other systems, is unknown. Human studies have shown that when a human has a salt appetite, the concentration at which they can detect the taste of salt reduces, they increase their preference for salty food, and they consume more salt.

When hyperaldosteronism is suspected in a hypertensive patient, they attend hospital for a day of investigations. Patient who are shown to have hyperaldosteronism have subsequent visits for imaging of their adrenals and sampling of blood from the adrenal vein to diagnose aldosterone producing adenomas (small tumours) which may be removed surgically, if not suitable for surgery, the hyperaldosteronism is treated with medication. This study will recruit hyperaldosteronism patients to investigate the effect of aldosterone on salt appetite by testing salt taste threshold, salt taste preference and intake before and after treatment.

DETAILED DESCRIPTION:
Aims

1. To determine if hypertensive patients with primary hyperaldosteronism have a lower salt taste threshold and heightened preference for salty soup compared to hypertensive patients with secondary aldosterone levels and a healthy control reference group.
2. To determine if treating primary hyperaldosteronism, with removal of aldosterone producing adrenal adenomas or medical blockade of aldosterone, results in changes in salt taste threshold and preference for salty soup.

   STUDY DESIGN

   This will be a non-interventional observational study examining a cohort of adult patients with hypertension under the care of Imperial College Healthcare NHS Trust who are being investigated and treated for primary hyperaldosteronism. No clinical intervention will occur as part of this study outside of their standard clinical practice. The schedule of events for each study will occur within 6 months.

   Visit 1 This coincides with the saline infusion test.

   According to the outcomes of the adrenal MDT discussion subsequent visits will depend on clinical plan (no further investigation or treatment, medical or surgical treatment) and will coincide with:

   Visit 2 i) adrenal venous sampling (to distinguish unilateral from bilateral disease). ii) clinic follow up after introduction of mineralocorticoid receptor antagonist (for patients deemed unsuitable for adrenal vein sampling)

   Visit 3 i) surgical outpatient assessment for removal of an adrenal adenoma. ii) clinic follow-up after introduction of mineralocorticoid receptor antagonists (for patients who carry unacceptably high risks for adrenal surgery or do not wish to have surgery, or deemed not suitable for removal of adrenal adenoma post adrenal vein sampling e.g. with bilateral disease).

   Visit 4 i) clinic follow up after adrenal adenoma removal.

   The protocol of investigation for each visit will consist of the following (total time ~60 mins ):

   Salt taste threshold testing This involves the participant, whilst blindfolded, tasting saline solutions, of varying concentration. The solution is sprayed onto the participant's tongue, the participant then states if the solution contains salt or not. Up to 20 solutions are tested (~10 mins) (Ohla et al., 2017).

   VAS and gLMS training Participants are trained to use labelled hedonic scales (LHS) (Wood et al., 2009) and general linear model sales (gLMS) (Green et al., 1996) to rate sensations using an established protocol (Veldhuizen et al., 2017) (5 mins) (Appendix 8).

   Salt taste preference testing This involves swilling a solution (soup of variable salt concentration) in the mouth then expectorating into a bowl. The subject then rates the solution on various parameters, for example liking, how it relates to "just right" saltiness, and intensity, using a gLMS. LHS or VAS. Each solution will be repeated 3 times. A sweet solution and bitter solution are also tested. This will take up to 40 mins.

   Saliva collection Saliva will be collected by asking participants to spit into a tube for up to 5 mins. Saliva will be analysed for electrolytes including sodium and potassium .

   Questionnaires i) Internal state questionnaire to assess internal state: hunger, thirst, fullness, pleasantness to eat, stress, anxiety, sleepiness, volume able to eat, nausea (5 mins) (Appendix 9).

   ii) Positive and Negative Affect Schedule (PANAS) to measure positive and negative mood (Watson et al., 1988).

   iii) Derby Salt questionnaire (DSQ) to assess habitual salt intake. iv) Beck's depression inventory (BDI) (visit 1 only) to screen for significant depression which is a contraindication

   3.3 Procedures

   3.3.1 Visit 1 (Saline infusion test) Patient arrives at 8 am (i) Blood pressure, heart rate, weight recorded on admission (standard care). (ii) Study explained, questions answered and patient is consented (iii) Patient is cannulated and blood taken for plasma aldosterone, plasma renin activity, U&Es (standard care).

   (iv) Patient remains in the seated position for at least 30 mins before infusion begins (standard care). During this time the taste tests are completed and saliva collected.

   (v) 2 litres of 0.9% saline are infused over 4 hours, starting at 9.00 a.m. (standard care). During this time the questionnaires will be completed.

   (vi) Blood pressure, oxygen saturation and heart rate are monitored throughout the test (standard care).

   (vii) After 4 hours (i.e. 1 pm), further blood sample are taken for aldosterone, renal function and electrolytes (standard care).

   (viii) Patient discharged as per standard clinical care.

   3.3.2 Visits 2-4 This will be dictated by clinical pathway according to outcome of the adrenal MDT discussion.

   3.3.2.1 Coincide with adrenal venous sampling. (i) Blood pressure, heart rate and weight recorded, and patient is cannulated on admission and blood samples sent (standard care).

   (ii) Confirmation is made that the patient is happy to continue with study. (v) Taste tests undertaken on the ward whilst the patient is waiting to go to the interventional radiology suite.

   (vi) Questionnaires will be completed if sufficient time. (vii) Adrenal venous sampling (standard clinical care) (viii) Post procedure observation period (standard clinical care). Questionnaires and taste tests completed if needed.

   (ix) Patient discharged after observation period (standard clinical care).

   3.3.2.2 Coincide with outpatient surgical consultation for adrenalectomy (If not convenient for the patient this may occur when the patient attends for pre-op assessment clinic).

   (i) Patient telephoned by the research team the week prior to appointment to remind the participant that study visit will occur and that the patient remains well.

   (ii) Patient attends clinic and has blood tests, observations and review by the surgical team, (standard care).

   (iii) Confirmation is made that the patient is happy to continue with study. (iv) Taste tests done and questionnaires will be completed in an out-patients room or Imperial NIHR Clinical Research Facility.

   3.3.2.3 Coincide with out-patient clinic follow-up visit after introduction of mineralocorticoid receptor antagonists or surgical removal of adrenal adenoma.

   (i) Patient telephoned by the research team the week prior to clinic appointment to remind the participant that study visit will occur and check that the patient remains well.

   (ii) Patient attends clinic and has blood tests, observations and review by endocrinology team (standard care).

   (iii) Taste tests done, saliva collected and questionnaires completed before or after clinical review in out-patients (Hammersmith, Charing Cross, St. Mary's Hospitals) or Imperial NIHR Clinical Research Facility, Hammersmith Hospital.

   (iv) Patient thanked for taking part in the study (this is the last visit).

   3.4 Saliva analysis and storage

   Saliva will be stored in the laboratories of Dr Tony Goldstone, PsychoNeuroEndocrinology Research Group. These are located in the, Commonwealth Building, Imperial College London, Hammersmith Hospital. This area has restricted access to research staff only and only research team members will have access to the stored samples. Following analysis samples will be stored by the research team pending ethical approval for use in another project.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Non-smoker (ex-smokers allowed)

Exclusion Criteria:

* Contra-indications for saline infusion test - severe uncontrolled hypertension, renal insufficiency, cardiac insufficiency, cardiac arrhythmia, or severe hypokalemia
* Current smoker
* Neurological disorder (moderate-severe traumatic brain injury, dementia)
* Significant current or past medical or psychiatric history, or use of medications, that, in the opinion of the Investigators, contraindicates their participation, due to influence on outcome measures.
* Patients lacking capacity or unable to consent
* Inability to understand verbal explanations or written information given in English
* Patients currently participating in an active CTIMP trial, or within 4 half-lives of last administration of CTIMP product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients with a raised plasma aldosterone/renin ratio being investigated for primary hyperaldosteronism.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Salt concentration taste threshold | 6 months
  Concentration of saline at which the salt taste is detected.
Ratings of salt liking and intensity across different salt concentrations | 6 months
  ratings of liking/wanting and intensity of soup containing differing concentrations of salt.

SECONDARY OUTCOMES:
Rating of sweet liking and intensity | 6 months
  ratings of liking/wanting and intensity of a sweet taste.
Rating of sour liking and intensity | 6 months
  rating of liking/wanting and intensity of a sour taste.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Salt taste thresholds. Taste ratings